CLINICAL TRIAL: NCT01105559
Title: Antibody Persistence in Healthy South African Children After Primary Series and Booster Vaccination With an Investigational (DTaP-IPV-Hep B-PRP-T) or Control Vaccines
Brief Title: Antibody Persistence in Healthy Children After Primary and Booster DTaP-IPV-Hep B-PRP-T Vaccine or Control Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: A3L26; UTN: U1111-1111-5789 (Other: WHO)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis
Keywords: Diphtheria; Tetanus; Whooping cough; Hepatitis B; Poliomyelitis; Diphtheria-Tetanus-acellular Pertussis Vaccines
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Participants previously received 3 doses and a booster dose of the investigational vaccine DTaP IPV Hep B PRP-T.
- Group 2: Participants previously received 3 doses CombAct-Hib™ + Engerix™ B + OPV and a booster dose of CombAct-Hib™ + Oral poliovirus vaccine (OPV) vaccine.
- Group 3: Participants previously received 3 doses DTaP IPV Hep B PRP-T; a dose of Engerix™ B at birth, and a booster dose of DTaP IPV Hep B PRP-T vaccine.

SUMMARY:
The purpose of this study is to evaluate the long term immunogenicity produced in children by the investigational hexavalent vaccine (DTaP-IPV-Hep B-PRP-T) given in Study A3L15 (NCT 00362336).

Primary Objective: To describe the antibody long term persistence at 3.5 and 4.5 years of age following a 3 dose primary series vaccination of either DTaP-IPV-Hep B-PRP-T or CombAct-Hib™ + Oral poliovirus vaccine (OPV) + Engerix™ B vaccination at 6, 10 and 14 weeks of age and a booster vaccination of DTaP-IPV-Hep B-PRP-T or CombAct-Hib™ + OPV at 15-18 months

DETAILED DESCRIPTION:
All participants must have received the primary series of vaccinations and a booster vaccination in Study A3L15 (NCT 00362336).

Participants will receive no vaccination in this study but will undergo immunologic assessments at 3.5 and 4.5 years of age.

ELIGIBILITY:
Inclusion Criteria :

* Aged 3 years and a half on the day of inclusion (42 months ± 60 days)
* Informed consent form signed by a parent or other legally acceptable representative and by an independent witness if the parent or other legal guardian is illiterate.
* Subject and parent/ legally acceptable representative able to attend the scheduled visits and to comply with all trial procedures.
* Receipt of primary vaccination with 3 doses of either DTaP-IPV-Hep B-PRP-T or CombAct-Hib™ + Oral poliovirus vaccine (OPV) + Engerix™ B and a booster dose of either DTaP-IPV-Hep B-PRP-T or CombAct-Hib™+ OPV.

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the inclusion in the trial.
* Incomplete primary and booster immunization at trial A3L15.
* Previous confirmed clinical, serological, or microbiological diagnosis of diphtheria, tetanus, whooping cough, poliomyelitis, Haemophilus influenza b or hepatitis B after completion of A3L15 Study.
* Subjects known to have received diphtheria, tetanus, pertussis, Haemophilus influenza b and hepatitis B vaccination after completion of A3L15 Study.
* Any vaccination within 30 days preceding inclusion, except for measles or poliovirus (monovalent) containing vaccines and pandemic influenza vaccines including pandemic H1N1-2009 strain, which may be received at least two weeks before the subject's blood sample collection
* Blood or blood-derived products received at the latest 3 months before inclusion, receipts of immunosuppressant drugs within the previous 3 months.
* Known or suspected congenital or acquired immunodeficiency since completion of A3L15 Study.
* Serious chronic illness occurring after receipt of the primary and booster series (e.g. leukemia, lymphoma [Tor B cells], Crohn's disease).
* Known or suspected subject seroconversion for human immunodeficiency virus (HIV) or hepatitis C seropositivity since completion of A3L15 Study.
* Febrile (temperature ≥ 38.0°C) or acute, moderate or severe systemic illness on the day of inclusion.

Ages: 41 Months to 43 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants aged 3 years and a half on the day of inclusion and must have received the primary series of vaccinations and a booster vaccination in Study A3L15 (NCT 00362336). No vaccination will be provided or administered in this study.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The antibody titers for each valence of DTaP-IPV-Hep B-PRP-T vaccine (except poliovirus) post-primary and booster vaccination. | Age 3.5 and 4.5 years after infant and booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- South Africa (2):
  - Bertsham
  - Johannesburg

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com